CLINICAL TRIAL: NCT02294201
Title: Spatial Repellent Products for the Control of Vector Borne Diseases - Malaria - Kenya
Acronym: SR-M-KEN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsors
Sponsor: University of Notre Dame (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SR-M-KEN
Record Dates: First submitted 2014-11-17; First posted 2014-11-19 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Malaria
Keywords: Malaria; Spatial Repellents; Plasmodium
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo Repellent product with no active ingredient
  Interventions: Device: Spatial Repellent product without active ingredient (SHIELD)
- Intervention (Active Comparator): Spatial Repellent product with active ingredient
  Interventions: Device: Spatial Repellent product with active ingredient; Device: Active ingredient

INTERVENTIONS:
Device: Spatial Repellent product with active ingredient — Spatial Repellent product
  Other Names: SHIELD
  Arms: Intervention
Device: Active ingredient — Transfluthrin (Active ingredient)
  Other Names: Transfluthrin
  Arms: Intervention
Device: Spatial Repellent product without active ingredient (SHIELD) — Spatial Repellent Product - Passive Emanator. The name of the product is SHIELD from SCJohnson
  Other Names: Placebo SHIELD
  Arms: Placebo

SUMMARY:
The primary objective of the study is to demonstrate and quantify the protective efficacy (PE) of spatial repellent products in reducing the incidence of malaria infection in human cohorts. The null hypothesis (H0) is that there is no difference in malaria incidence between intervention and control arms.

DETAILED DESCRIPTION:
The primary epidemiological endpoint will be the incidence density of first time malaria infections among human cohorts during the follow-up period as detected by polymerase chain reaction assay (PCR). This measure will inform PE (the reduction of incidence) between intervention and control study arms using the formula: PE =[(Ip - Ia)/Ip]* 100%; based on an expected minimum effect size of 30%. First time infections in these subjects will offer relatively unambiguous evidence of the extent of exposure to infectious mosquito bites. The primary entomological endpoint will be adult densities of vector species via human-landing catch (HLC) from sentinel households from intervention and control arms over the follow-up period.

Secondary epidemiological endpoints will be the incidence density of first time malaria infections among human cohorts during the follow-up period as detected by microscopy and the total number of cases averted (i.e., all Plasmodium spp. infections in cohort subjects). Secondary entomological endpoints include number of sporozoite infected mosquitoes, parity and species-specific effects of the spatial repellent product.

Both epidemiological and entomological endpoints will be utilized to look at the relationship between SR and PE based on product coverage (to include diversion and community effects) and insect behavior. The prospect of SR associated temporal cumulative effects on study endpoints (epidemiological and entomological) over transmission seasons will also be investigated by using the cumulative incidence of infection over the season and applying a survival curve analysis of the cohort data.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-59 months
* glucose-6-phosphate dehydrogenase (G6PD) normal (qualitative screen) in sites where P. vivax or P. ovale known prevalence rates represent major burden) and whose treatment with primaquine is implemented within national guidelines
* Hb > 5mg/dl
* Temperature ≤38.0°C) and no moderate or severe acute illness/infection on the day of inclusion
* Sleeps in cluster >90% of nights during any given month
* No plans for extended travel (<1month) outside of home during study
* Not participating in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure during the trial
* Provision of assent/informed consent form signed by the subject and by the parent(s) or another legally acceptable representative

Exclusion Criteria:

* children < 6 months or > 5 years
* G6PD deficiency (qualitative screen) in sites where P. vivax or P. ovale known prevalence rates represent major burden and whose treatment with primaquine is implemented within national guidelines
* Severe anemia
* Febrile illness (temperature ≥38.0°C) or moderate or severe acute illness/infection on the day of inclusion
* Sleeps in cluster <90% of nights during any given month
* Plans for extended travel (>1month) outside of home during study
* Participating or planned participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure during the trial
* No provision of assent/informed consent form signed by the subject and by the parent(s) or another legally acceptable representative

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Malaria Incidence | 104 weeks
  Incidence of malaria infections among human cohorts during the follow-up period as detected by PCR

CONTACTS AND LOCATIONS:
Overall Officials: Neil Lobo, PhD, Principal Investigator — University of Notre Dame; Nicole Achee, PhD, Principal Investigator — University of Notre Dame
Locations (1):
- Kemri-Crc, Kisumu, Kenya